CLINICAL TRIAL: NCT03561116
Title: Effects of Xanthohumol on Metabolic Syndrome Progression (XAN4Health)
Brief Title: Effects of Xanthohumol on Metabolic Syndrome Progression
Acronym: XAN4Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XAN4Health
Record Dates: First submitted 2018-05-24; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Xanthohumol; Glucose metabolism; DNA damage
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XAN (Experimental): XAN (1 sachet of 12 mg/day)
  Interventions: Dietary Supplement: XAN
- Placebo (Placebo Comparator): Placebo (1 sachet with excipient)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: XAN — Daily intake of a sachet containing 12 mg of XAN
  Arms: XAN
Dietary Supplement: Placebo — Daily intake of a sachet containing excipient
  Arms: Placebo

SUMMARY:
A huge body of scientific evidence has suggested that xanthohumol (XAN) consumption, a polyphenol present in beer, has a positive effect on energy metabolism. This compound is known for its antioxidant, anti-inflammatory and anti-cancer properties which confer potential to be used as a food supplement. Nevertheless, XAN lipophilic properties prevent the extensive use of this molecule as a functional food compound. The company TA-XAN S.A.M. (Wiesbaden, Germany) has patented a method to overcome this solubility problem. So, the main aim of this study is to evaluate the effects of XAN consumption on metabolic syndrome progression in individuals recently diagnosed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 25-65 years of age;
* Criteria for metabolic syndrome according to the 2005 revised NCEP ATP III guidelines:

  * HDL-C < 40 mg/dL ♂ and < 50 mg/dL ♀;
  * Triglycerides ≥ 150 mg/dL;
  * Blood pressure ≥ 130/85 mmHg;
  * Fasting plasma glucose ≥ 100 mg/dL;
  * Waist circumference ≥ 102 cm ♂ and ≥ 88 cm ♀;
* HbA1c 5.8/6.0-6.4;
* Nonsmokers or no other tobacco use in the last 3 months;
* Willing to stop taking regular supplements including antioxidants for 2 weeks prior to study entry through conclusion of study;
* Willing to stop consumption of beer for 2 weeks prior to study entry through conclusion of study;
* Must be able to provide informed consent;
* Blood screen tests [comprehensive metabolic panel (CMP), and lipid profile] within normal limits or if outside normal limits, approved for participation at the discretion of the study physician.

Exclusion Criteria:

* Have a significant acute or chronic coexisting illness, such as cardiovascular disease, chronic kidney or liver disease, gastrointestinal disorder, endocrine disorder, immunological disorder, metabolic disease, cancer, chemotherapy history, gluten intolerance, eating disorders, depression or any psychiatric condition, diabetes, or any condition which contraindicates entry in the study, according to the investigators' judgment;
* Currently taking prescription drugs other than oral contraceptives (over-the-counter medications are allowed upon review and discretion of the study physician);
* Consumption of more than the recommended alcohol guidelines (> 1 drink/day ♀ and > 2 drinks/day ♂);
* Consumption of high levels of beer;
* Pregnancy (as confirmed by urine pregnancy test) or planning to become pregnant before completing the study;
* Breastfeeding;
* Under UV therapy (e.g. psoriasis treatment), using UV tanning beds and unprotected sun exposure greater than 1 hour/day;
* Engaging in vigorous exercise more than 6 hours/week;
* Participation in other dietary study in the past 3 months;
* Had surgery in the last 3 months;
* Post-menopausal status.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-05-19 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | Change from baseline of HbA1c at 3 months
Comet assay | Change from baseline of DNA damage at 3 months

SECONDARY OUTCOMES:
HDL-cholesterol | Change from baseline of HDL-cholesterol at 3 months
LDL-cholesterol | Change from baseline of LDL-cholesterol at 3 months
Triglycerides | Change from baseline of triglycerides at 3 months
Total-cholesterol | Change from baseline of total-cholesterol at 3 months
Waist circumference | Change from baseline of waist circumference at 3 months
Body weight | Change from baseline of body weight at 3 months
Body composition | Change from baseline of body composition at 3 months
Blood pressure | Change from baseline of blood pressure at 3 months
Heart rate | Change from baseline of heart rate at 3 months
ApoB | Change from baseline of ApoB at 3 months
ApoA1 | Change from baseline of ApoA1 at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Soares, PhD, Principal Investigator — Medical Faculty of University of Porto
Locations (1):
- Medical Faculty of University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided